CLINICAL TRIAL: NCT01172574
Title: Motor Control Exercise Can Reduce Pain and Improve Postural Alignment in Osteoporotic Women With Vertebral Fractures: a Randomized Controlled Trial
Brief Title: Motor Control Exercise in Osteoporotic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Dr. Palina Karakasidou, Researcher, Laboratory for Research of the Musculoskeletal System, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1112
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2008-01

CONDITIONS: Osteoporosis; Postmenopausal
Keywords: Osteoporosis; Pain; Kyphosis; Posture; Exercise therapy
MeSH Terms: conditions — Osteoporosis; Pain; Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motor control exercise (Experimental): Subjects of the exercise group underwent a 3-month (13-week) treatment program directed on 3-weekly 1-hr one-to-one sessions by the researcher who had experience in the specific exercise treatment of the spinal region. During the next 3 months, the subjects were urged to perform the exercises alone at home at least once a day, and compliance was monitored by the activity quota chart given to them at the beginning of each study-month.
  Interventions: Other: Motor control exercise
- Control group (No Intervention): The control group underwent treatment throughout a 6-month period, directed by each patient's medical practitioner. This consisted of the patients carrying out regular weekly general exercises (walking and swimming). Three of them regularly attended other treatment providers involving group general exercise programs. Two patients received the application of local pain-relieving methods such as heat, massage, laser and ultrasound and one did nothing except for receiving osteoporotic medication.

INTERVENTIONS:
Other: Motor control exercise — Participants of the exercise group were trained to consciously co-activate the transversus abdominis, pelvic floor and thoracic erector spinae muscle, relax the lumbar multifidus and use the diaphragmatic breathing pattern. They were encouraged to activate the specific muscles of the trunk regularly during daily activities, particularly in situations where they anticipated or experienced pain such as walking, twisting, lifting low-lying objects and working with the hands in sitting or standing positions
  Arms: Motor control exercise

SUMMARY:
The objective of this study was to explore the effectiveness of Motor Control Exercise on pain, postural alignment and spinal curvatures in women with osteoporotic vertebral fractures.

DETAILED DESCRIPTION:
Osteoporosis is a common metabolic bone disease that usually affects the aging population. It is an important public health problem, due to its association with vertebral and nonvertebral fractures leading to increased morbidity. Vertebral fractures are accompanied by kyphosis, reduced pulmonary function, loss of height, and are often associated with elevated pain while they may also lead to subsequent vertebral fractures. Osteoporotic individuals exhibit kyphosis in the erect standing position, which, in turn, is compensated by the deformation of other parts of the body. Improvement of postural alignment may lead to less stress on the spine, facilitate posture and proper body mechanics and may improve balance. The aim of the present study was to assess the effectiveness of Motor Control Exercise on pain, postural alignment and spinal curvatures in women with osteoporotic vertebral fracture against the results of a control group that received the basic therapies for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporosis
* Osteoporotic vertebral fractures
* Pain
* Under medical osteoporotic treatment

Exclusion Criteria:

* osteoporosis other than primary postmenopausal
* vertebral collapse with neurological deficits
* more than 5 fractured vertebrae
* major respiratory conditions
* receiving pain reducing agents, teriparatide or calcitonin

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pain | Baseline
  Pain was assessed using the visual analogue scale (VAS) of 11 numerical points (0='no pain', 10='worst imaginable pain'). Participants were asked to verbalize the presence of pain in their trunk and lower limbs during the previous 2 weeks.
Pain | 3 months
  As described
Pain | 6 months
  As described

SECONDARY OUTCOMES:
Photographic measurements | Baseline
  Two-dimensional posture photography was performed using a digital Video Camera. With participants in their underwear, self-adhesive patches of 1.5 cm were placed over the left-side lateral landmarks. Women were instructed to stand in a comfortable posture with feet 20 cm apart. The participants were photographed twice at each time point. The photographs were analyzed by measuring the angles between a perpendicular line transcending the lateral malleolus, head of fibula, great trochanter, shoulder and ear. The mean of each angle of both photographs was used for statistical analysis.
Spinal curvatures | Baseline
  These were measured using a Sounders digital inclinometer according to the instruction manual. Standing thoracic, lumbar, and lumbosacral angle were measured. The examiner repeated the procedure three times, and if the measurements differed by more than 5 degrees, they were repeated and the second set of measurements recorded.
Photographic measurements | 3 months
  As described
Spinal curvatures | 3 months
  As described
Photographic measurements | 6 months
  As described
Spinal curvatures | 6 month
  As described

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Thias Pronoias 'I Pammakaristos', Athens, Attica, Greece